CLINICAL TRIAL: NCT00164034
Title: Trauma Reception and Resuscitation Project - 'Time for a New Approach'
Brief Title: Trauma Reception and Resuscitation Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: Victorian Trauma Foundation (Other); National Trauma Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 166/03
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2005-09

CONDITIONS: Trauma
Keywords: Trauma; Wounds; Injuries
MeSH Terms: conditions — Wounds and Injuries

INTERVENTIONS:
Device: Real time computer prompted trauma algorithms

SUMMARY:
Test the hypothesis that the implementation of real-time, computer-prompted algorithms in the first half hour of trauma management will result in a measurable reduction in management errors associated with the reception and resuscitation of major trauma patients.

Demonstrate that a reduction in management errors will translate into a reduction in morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria: All injured patients > 15 years old who are brought or present to the The Alfred Trauma Centre during the study period.

Exclusion Criteria: Stable Trauma patients (ie Pulse rate <100/minute, MAP >70mmHg, Hb >70, temperature >35 and <37.5, Spo2 >92%, GCS >13) undergoing secondary transfer from another hospital, where trauma occurred >6hrs prior to arrival.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1171 (Actual)
Dates: Start 2005-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Error rate per patient treated demonstrated by deviation from the algorithms

SECONDARY OUTCOMES:
Missed injuries
Time to decision

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fitzgerald, MBBS, FACEM, MRCMA, Principal Investigator — The Alfred Hospital, Bayside Health, Melbourne, Australia
Locations (1):
- The Alfred Hospital, Emergency and Trauma Centre, ., Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Fitzgerald M, Cameron P, Mackenzie C, Farrow N, Scicluna P, Gocentas R, Bystrzycki A, Lee G, O'Reilly G, Andrianopoulos N, Dziukas L, Cooper DJ, Silvers A, Mori A, Murray A, Smith S, Xiao Y, Stub D, McDermott FT, Rosenfeld JV. Trauma resuscitation errors and computer-assisted decision support. Arch Surg. 2011 Feb;146(2):218-25. doi: 10.1001/archsurg.2010.333. PMID 21339436
- See also: National Trauma Research Institute — http://www.ntri.org.au/
- See also: The Alfred Hospital, Melbourne, Victoria, Australia. — http://www.alfred.org.au